CLINICAL TRIAL: NCT06246240
Title: Effect of Vitamin C Chewing Gum on Pregnancy Nausea and Vomiting Severity: Randomized Controlled Study
Brief Title: Vitamin C Chewing Gum, Pregnancy Nausea and Vomiting
Acronym: PregnancyNause
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Fatma Yildirim, Dr., Hitit University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: Hitituniversity_1
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Pregnancy Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Chewing Gum; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The Personal Information Form will be applied to the control group without any intervention and they will be asked to score the VAS Scale at the time the nausea begins and the retests at 60 and 120 minutes. After the interview with the pregnant women, all pregnant women will be called 24-48 hours later and data will be collected by questioning the 60th and 120th minute VAS scores of nausea severity.
- Intervention group (Experimental): After obtaining the consent of the pregnant women, the Personal Information Form and VAS scale were applied. The experimental group was asked to score the VAS scale as soon as nausea started and was practiced chewing vitamin C gum for 30-60 minutes. Pregnant women in the experimental group were asked to score the VAS scale at 60 and 120 minutes after chewing gum.
  Interventions: Other: Chewing gum with vitamin C

INTERVENTIONS:
Other: Chewing gum with vitamin C — Will chew vitamin C gum as soon as nausea begins
  Arms: Intervention group

SUMMARY:
Although there are studies in the literature examining the effects of chewing gum or using vitamin C on nausea and vomiting symptoms, no study has been found examining the effect of vitamin C gum on the severity of nausea and vomiting during pregnancy. This study aimed to investigate the effect of vitamin C gum on the severity of pregnancy nausea and vomiting.

DETAILED DESCRIPTION:
One of the problems that occur during pregnancy, the etiology of which is not fully known, is nausea and vomiting experienced during early pregnancy (Taşkın, 2019). Meta-analysis studies indicate that the prevalence of nausea and vomiting during pregnancy is between 35% and 91% (Matthews et al., 2015; Sridharan and Sivaramakrishnan, 2018). Nausea and vomiting usually occur on days 4-6. It starts in weeks 9-16 of pregnancy. It peaks in the following weeks (Matthews et al., 2015). Risk factors for nausea and vomiting during pregnancy are not known precisely. While the increase in human chorionic gonadotropin hormone and estrogens in the blood seems to be the possible cause, hormonal factors such as prostaglandin E2, thyroxine and prolactin are probably added to this (Bustos et al., 2017). There are many pharmacological and non-pharmacological methods with proven effects in the treatment of pregnancy nausea and vomiting. Pharmacological treatments include antiemetics, anticholinergics, antihistamines, dopamine antagonists, vitamins (B6 and B12), H3 antagonists or combinations of these substances (Erişen et al., 2021). Non-pharmacological methods include some interventions such as acustimulation, acupuncture, chamomile, ginger, peppermint oil, lemon oil, and vitamin B6 (Matthews et al., 2015). Pregnant women with nausea and vomiting generally do not want to receive pharmacological treatment due to concerns about the negative effects of drugs on the fetus. It is stated that various vitamin-based products such as B6, B12 and herbal treatments such as ginger, mint, peppermint oil and lemon are effective and safe in pregnancy nausea and vomiting (Sarecka-Hujar and Szulc-Musioł, 2022).

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* At least primary school graduate,
* married,
* Those who are younger than the 16th week of pregnancy,
* Those who complain of nausea and vomiting during pregnancy,
* Those who agreed to participate in the study.

Exclusion Criteria:

* Those who have a health problem that may cause nausea and vomiting in their current pregnancy,
* Those receiving any antiemetic treatment,
* Smokers.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 78 (Estimated)
Dates: Start 2023-10-08 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-03-05 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 0-60-120. munites
  It will be used to measure the severity of nausea and vomiting.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatma Yıldırım, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided